CLINICAL TRIAL: NCT03772418
Title: Formulation and Evaluation of Topical Preparation Containing Pomegranate and Ginkgo Biloba for Anti-aging Activities
Brief Title: Topical Preparation of Pomegranate and Ginkgo Biloba for Anti-aging Activities
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed A. H. Abdellatif (Other)
Responsible Party: Sponsor-Investigator, Ahmed A. H. Abdellatif, Assistant Prof. at Pharmaceutics dept., Faculty of Pharmacy, Qassim University, KSA, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharPGB
Record Dates: First submitted 2018-05-15; First posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Skin and Subcutaneous Tissue Disorders
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cream base (Placebo Comparator): A group of volunteers receiving placebo medications without natural extracts of ginkgo biloba and Pomegranate.
  Interventions: Drug: Cream Base
- Pomegrante and Ginkgo biloba group (Active Comparator): A group of volunteers with the aging state receiving natural extracts of ginkgo biloba and Pomegranate in different topical dosage forms.
  Interventions: Drug: Pomegrante and Ginkgo biloba group

INTERVENTIONS:
Drug: Cream Base — The formulated dosage form without ginkgo biloba or pomegranate will be applied to the 30 aging people who are suffering from wrinkles in the skin male and female. Typically, will be applied on two groups, one man (Group 0a) and one woman were (Group 0b) which they will be used plain cream.
  Other Names: Aging group recieving placebo dosage form
  Arms: Cream base
Drug: Pomegrante and Ginkgo biloba group — The extracts of ginkgo biloba and Pomegranate as formulated in topical dosage form will be applied to the 30 aging people who are suffering from wrinkles in the skin male and female. Formulated cream will be applied on two groups, one man (Group Ia)and one woman (Group Ib).
  Other Names: Aging group receive ginkgo biloba and Pomegranate
  Arms: Pomegrante and Ginkgo biloba group

SUMMARY:
As the quality of life improves, people are seeking to look as young as they feel. Ginkgo biloba (GB) and Pomegranate (PG) extract can be used to create efficacious topical anti-aging products. GB & PG are now widely used in research and clinical trials on age-associated diseases, for example, skin aging, brain dysfunction, cardiovascular system diseases, carcinogen metabolism. The investigator's aim is to formulate a topical cream in the form (O/W or W/O emulsion) formulation, containing GB as an anti-aging formulation for the public.

DETAILED DESCRIPTION:
In this study, a vanishing cream will be prepared by reaction of a stearic acid with alkali (NaOH) to form stearate soap. Then the GB extract will be added to the final form. The formulated cream will be characterized for identifying the type of emulsion, calibration curve for GB, drug content, irritation to skin, homogeneity test, pH, FT-IR test, ex vivo studies, physical stability, and human application. Finally, a 9-questions questionnaire was published using Google forms for the human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of aging shape
* Follow up and collect data for a local and systemic activity of Ginkgo Biloba and Pomegranate
* The skin should be not injured as the cream can be easily applied
* Systemic oral capsule Ginkgo Biloba and Pomegranate can be also given to enhance the activity as anti-aging activity

Exclusion Criteria:

* Insulin-dependent diabetes
* Hypertension disease
* Skin wound

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of ant-aging activity of Pomegranate and Ginkgo biloba | Three months
  The crow's feet wrinkle of 17 volunteers will be measured compared to the control group. The significant results will measure the decrease in the depths of deep furrows for groups treated with Pomegranate and Ginkgo biloba over a three months period.

SECONDARY OUTCOMES:
Stable topical anti-aging products for long life shelf storage | Six months
  Stability test will be studied for dosage forms. The test will be carried out by standing the products on shelf life for six months. The stability test will be recorded using high-performance liquid chromatography each thee days.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdellatif, Ph.D., Principal Investigator — Assistant Prof. at Pharmaceutics dept., Faculty of Pharmacy, Qassim University, KSA
Locations (3):
- Assiut Clinic, Asyut, Egypt
- Saudi Arabia (2):
  - Faculty of Pharmacy, Buraidah, Al-Qassim Region
  - Pharmaceutics dept., Faculty of Pharmacy, Qassim University, Buraidah, Al-Qassim Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dong LY, Fan L, Li GF, Guo Y, Pan J, Chen ZW. [Anti-aging action of the total lactones of ginkgo on aging mice]. Yao Xue Xue Bao. 2004 Mar;39(3):176-9. Chinese. PMID 15171650
- [Background] Kang SJ, Choi BR, Kim SH, Yi HY, Park HR, Song CH, Ku SK, Lee YJ. Beneficial effects of dried pomegranate juice concentrated powder on ultraviolet B-induced skin photoaging in hairless mice. Exp Ther Med. 2017 Aug;14(2):1023-1036. doi: 10.3892/etm.2017.4626. Epub 2017 Jun 16. PMID 28810554
- [Result] Rasul A, Akhtar N. Formulation and in vivo evaluation for anti-aging effects of an emulsion containing basil extract using non- invasive biophysical techniques. Daru. 2011;19(5):344-50. PMID 22615680